CLINICAL TRIAL: NCT02211911
Title: Investigation of the Pharmacokinetics of 10 mg Bisacodyl (Coated Tablets) or 10 mg Sodium Picosulfate (Drops) Administered Orally in Healthy Lactating Females
Brief Title: Pharmacokinetics of Bisacodyl or Sodium Picosulfate Administered Orally in Healthy Lactating Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122.57
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Bisacodyl; picosulfate sodium

ARMS (2):
- Bisacodyl (Experimental)
  Interventions: Drug: Bisacodyl
- Sodium picosulfate (Experimental)
  Interventions: Drug: Sodium picosulfate

INTERVENTIONS:
Drug: Bisacodyl
  Arms: Bisacodyl
Drug: Sodium picosulfate
  Arms: Sodium picosulfate

SUMMARY:
To investigate if bisacodyl (Dulcolax®) and sodium picosulfate (Laxoberal®) is excreted in breast milk of healthy lactating women after an oral administration of 10 mg once daily over a period of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Women, age ≥18 and ≤50 years
* Stopped with breast feeding their baby
* Provided breast milk samples over a period of 10 days (including day -1)
* Have been breast feeding for at least 14 days
* Complied with the requirements of the protocol (e.g complete a diary)
* Body Mass Index (BMI) ≤ 35 kg/m2
* Medically acceptable method of contraception [i.e., double barrier method (e.g., diaphragm or condom and spermicide), hormonal therapy (subcutaneous, injectable, intra-vaginal, or oral contraceptive) or intrauterine device
* Signed and dated a written informed consent prior to any study procedures study in accordance with Good Clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Findings during medical examination (including BP, pulse rate and ECG) deviating from normal and of clinical relevance
* Evidence of clinically relevant concomitant diseases like renal insufficiency, cardiac insufficiency, myocardial infarction, other known cardiovascular disease including hypertension
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, that may interfere with the safety of the subject
* Surgery of the gastrointestinal tract (except appendectomy) in the last 2 years
* Metabolic disorders, neurological disorders, severe or psychiatric disorders, or any other significant disease or intercurrent illness (e.g. abdominal/gastrointestinal surgery) that would interfere with participation in the study
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. HIV, Hepatitis)
* Participated in another study with an investigational product within 1 month prior to enrolment into this study or during the study
* Eating disorder
* Hypersensitivity to bisacodyl, sodium picosulfate or any of the inactive ingredients
* Any concomitant medication except for paracetamol or hormonal therapy.
* Abnormal electrolyte values at the screening visit. The electrolyte values should be within the normal ranges
* Alcohol abuse; subjects who report regular consumption of 40g/day = 5 units/day or more alcoholic drinks per day were excluded
* Smoker (>10 cigarettes or > 3 cigars or > 3 pipes/day)
* Drug abuse
* Any laboratory value outside the reference range that is of clinical relevance
* Mastitis
* Less than 200 ml daily (24 hours) production of breast milk on day -1
* A positive pregnancy test at screening

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 8 days
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | up to 8 days
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose) | up to 8 days
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 8 days
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable concentration at tz) | up to 8 days
%AUCtz-∞ (the percentage of the AUC 0-∞ that is obtained by extrapolation) | up to 8 days
λz (terminal rate constant in plasma) | up to 8 days
t1/2 (terminal half-life of the analyte in plasma) | up to 8 days
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 8 days
CL/F (apparent clearance of the analyte in plasma following extravascular administration) | up to 8 days
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular administration) | up to 8 days
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | up to 8 days
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 8 days
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 8 days
Aet1-t2,milk (amount of analyte in milk from the time point t1 to time point t2) | up to 8 days
fet1-t2,milk (fraction of analyte in milk from time point t1 to time point t2) | up to 8 days
AUCτ,milk (area under the concentration-time curve of the analyte in milk over a uniform dosing interval τ after administration of the first dose) | up to 8 days
milk to plasma ratio (AUCτ,milk / AUCτ) | up to 8 days
estimated daily infant dosage | up to 8 days
  (milk-to-plasma ratio x average maternal plasma concentration x 150 mL/kg/day)
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 8 days

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 8 days
Number of patients with abnormal laboratory findings | up to 8 days
Number of patients with abnormal electrocardiogram findings | up to 8 days
Number of patients with clinically significant changes in vital signs | up to 8 days
Number of bowel movements | up to 8 days